CLINICAL TRIAL: NCT05264831
Title: Pulmonary Vein Isolation Alone or in Combination With Substrate Modulation After Electric Cardioversion Failure in Patients With Persistent Atrial Fibrillation: a Randomized, Multicentric, and Comparative Study
Brief Title: Pulmonary Vein Isolation Alone or in Combination With Substrate Modulation After Electric Cardioversion Failure
Acronym: PACIFIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PACIFIC; 2021-A02291-40 (Other: ANSM)
Record Dates: First submitted 2022-02-03; First posted 2022-03-03 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Single Person

STUDY DESIGN:
Intervention Model Description: The study procedure is the electric cardioversion as a discriminant factor between patients requiring PVI procedure alone or PVI procedure combined with substrate modulation. This electric cardioversion will be performed in all included patients up to 6 weeks before the ablative procedure.
  On the day of the ablative procedure:
  * If the patient presents with a Sinus Rhythm (= successful electric cardioversion, approximately 70% of patients) the patient will be treated as per SoC in accordance with ESC recommendations. It is recommended to perform PVI procedure alone in these patients. A prospective registry for these patients will be established for this study.
  * If the patient presents with AF (= failure of electric cardioversion, approximately 30% of patients), randomization will be carried out according to the 2 strategies:
  * Group 1: PVI procedure alone in accordance with ESC recommendations
  * Group 2: PVI procedure associated with substrate modulation
Masking Description: N/A, open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVI procedure alone (Active Comparator): If the patient presents with AF (= failure of electric cardioversion, approximately 30% of patients), randomization will be carried out according to :
  - Group 1: PVI procedure alone in accordance with ESC recommendations
  Interventions: Procedure: Pulmonary Vein Isolation (PVI) alone
- PVI procedure combined with substrate modulation (Experimental): If the patient presents with AF (= failure of electric cardioversion, approximately 30% of patients), randomization will be carried out according to :
  - Group 2: PVI procedure associated with substrate modulation
  Interventions: Procedure: PVI procedure associated with substrate modulation

INTERVENTIONS:
Procedure: Pulmonary Vein Isolation (PVI) alone — PVI procedures correspond to point-by-point 50W AI-guided RF applications (400 posterior LA wall, and 550 elsewhere). The PVI will be validated by the absence of any activity recorded inside the PV encirclement by a multipolar catheter (either a Lasso catheter or a Pentaray catheter) (entrance block) and by the non-capture of the LA despite pacing maneuvers from inside the encirclement (exit block). The bidirectional block will be validated again after a 15-minutes waiting period.
  Arms: PVI procedure alone
Procedure: PVI procedure associated with substrate modulation — PVI procedure associated with substrate modulation
  Arms: PVI procedure combined with substrate modulation

SUMMARY:
This study aims at assessing whether electric cardioversion can act as a discriminant factor between patients requiring Pulmonary Vein Isolation (PVI) procedure alone or PVI procedure combined with substrate modulation.

All included patients will undergo an electric cardioversion, then:

* Patients with electric cardioversion success will be treated as per Standard of Care and according to ESC recommendations (2020). A prospective registry will be implemented for these patients.
* Patients with electric cardioversion failure will be randomized in the study between 2 ablative procedures:

  * PVI procedure alone
  * PVI procedure combined with substrate modulation

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common heart rhythm disorder. It is the result of uncoordinated action of the atrial myocardial cells, causing rapid and irregular contraction of the heart's atria.

The AF prevalence in adults is currently estimated to be between 2% and 4% and is expected to increase by a factor of 2.3 in the next few years, due to the increased longevity of the general population and the increased search for undiagnosed AF. Increased age is an important risk factor for AF, but other increased comorbidities, including hypertension, diabetes, heart failure, coronary artery disease, chronic renal failure, obesity, and obstructive sleep apnoea syndrome, are also important; modifiable risk factors contribute strongly to the development and progression of AF (ESC Guideline, 2020).

The European Society of Cardiology (ESC) recommended pulmonary vein isolation (PVI) (Class IA) as first-line ablative strategy for persistent AF (Class IA) (ESC Guideline, 2020). However, PVI alone is only effective in treating about 40% to 60% of patients with persistent AF in the general population (unselected). If we apply this strategy to all patients (PVI alone), we accept to re-do ablative procedure in up to 60% of patients.

The second feasible strategy is to treat patients with persistent AF by PVI combined with substrate modulation (ESC Class IIb). This strategy, when done well, by creating irreversible lesions (Marshall-PLAN) can effectively treat 70% to 80% of AF patients. But this implies that the investigator will be doing unnecessary substrate modulation in up to 40% of patients, which can lead to increased risks associated with the ablative procedure, longer procedure times, multiple lesions, etc… In addition, incorrect or incomplete substrate modulation is pro-arrhythmic and leads to recurrences in the form of left atrial flutters, tolerance of which, is generally poor.

Both ablative strategies have been widely validated in large numbers of published studies.

The problem is to know when and for which patients to apply one or the other of the two strategies. Electric cardioversion could help in selecting the most appropriate strategy.

ELIGIBILITY:
Inclusion criteria:

Criteria to be validated for patients included before performing electric cardioversion:

1) Persistent AF (continuous for at least 7 days without interruption according to information transmitted by the cardiologist and the patient), symptomatic and resistant to at leat one anti-arrhythmic drug treatment including amiodarone;

Criteria to be validated for patients included after performing electric cardioversion :

1. Patient treated by electric cardioversion for persistent AF, symptomatic and resistant to anti-arrhythmic treatment including amiodarone and whom ablative procedure is planned in the following 4-6 weeks after electric cardioversion

   Criteria to be validated for all patients included:
2. Life expectancy > 5 years;
3. Female or male between 18 and 80 years of age at the electric cardioversion time
4. Affiliation to a health insurance system;
5. Patient informed of the study and having signed informed consent

   Criteria to be validated prior to randomization on the day of ablation (these patients may be randomized):
6. Patient with failed electric cardioversion i.e. in AF, confirmed by ECG.

Exclusion criteria:

Criteria to be validated before or after performing electric cardioversion (the study cannot be proposed to patients corresponding to these criteria):

1. Current hyperthyroidism;
2. Pregnant or breastfeeding woman;
3. Patient with a Body Mass Index (BMI) greater than 35;
4. Patient with severe Chronic Obstructive Pulmonary Disease (COPD);
5. Patient with hypertrophic heart disease;
6. Patient with a mechanical or biological mitral valve;
7. Contraindications to anticoagulants;
8. Transient Ischemic Attack (TIA) /stroke less than 6 months old;
9. Psychiatric illness affecting follow-up;
10. Left Ventricular Ejection Fraction (LVEF) < 40% ;
11. Uncontrolled ischaemic heart disease (angina, myocardial ischaemia)
12. Patients under legal protection
13. Cardiac surgery on left atrium
14. Inflammatory status in progress (cancer, rheumatoid arthritis, PPRZ, acute or chronic periodontitis, Crohn's disease, RCUH)
15. Pulmonary embolism or phlebitis less than 6 months old
16. Prior atrial fibrillation ablation
17. Active cancer

    Criteria to be validated before randomization, on the day of ablation (these patients cannot be randomized):
18. Patient in sinus rhythm 4-6 weeks after electric cardioversion: these patients are included in the study registry.
19. Patient with complete absence of sinus rhythm (less than 10 seconds) after 3 electric cardioversion attempts: these patients will discontinue from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
1-year sinus rhythm maintenance rate | At 1 year after ablation
  Rate of patients with sinus rhythm (yes/no) at 1 year after a single ablative procedure

SECONDARY OUTCOMES:
Rate of patients with sinus rhythm (randomized patients) | At 1 year after ablation
  Rate of patients with sinus rhythm during 1 year after ablation and after a single ablative procedure.
Rate of patients with sinus rhythm (registry patients) | At 1 year after ablation
  Rate of patients with sinus rhythm during 1 year after ablation and after a single ablative procedure.
Rate of patients with sinus rhythm (randomized and registry patients, strategy PVI procedure alone) | At 1 year after ablation
  Rate of patients with sinus rhythm during 1 year after ablation and after a single ablative procedure.
Duration (in minutes) of ablative procedure | On the day of the ablative procedure
  Duration (in minutes) of ablative procedure
Duration (in minutes) of radiofrequency use | On the day of the ablative procedure
  Duration (in minutes) of radiofrequency use
Duration (in minutes) of Fluoroscopy | On the day of the ablative procedure
  Duration (in minutes) of Fluoroscopy
Duration (in days) of hospitalization | From date of surgery until the date of discharge from hospital assessed up to 1 day
  Duration (in days) of hospitalization
Evaluation of major complications rate | Up to 1 year
  Tamponade and/or stroke rate out of the blanking period and up to 1-year follow-up
Evaluation of drug treatment use rate or electric cardioversion in the blanking period | At three months after ablation
  Number of patients using drug treatment and/or electric cardioversion during the blanking period (first 3 months after ablation) between the two strategies (randomized patients)
Evaluation of the minor complications rate between the two strategies after 1-year follow-up (randomized patients) | up to 1-year follow-up
  Occurrence of a false aneurysm or fistulas at the puncture sites and/or occurrence of a post-ablation pericardial reaction
Evaluation of the vein isolation as well as other linear lesions in patients with recurrence of atrial fibrillation during 1 year after ablation | up to 1-year follow-up
  Pulmonary vein isolation as well as other linear lesions block assessment during redo procedures
Evaluation of the impact of low voltage areas on the response to EC prior to catheter ablation | catheter ablation
  Relationship between the presence or absence of LA low voltage areas and the response to EC prior to catheter ablation Relationship between the extent of LA low voltage areas and the response to EC prior to catheter ablation Relationship between the location of LA low voltage areas and the response to EC prior to catheter ablation
Evaluation of the impact of low voltage areas on the success of the ablation procedure | ablation procedure
  Relationship between the presence or absence of LA low voltage areas and the success of the ablation procedure Relationship between the extent of LA low voltage areas and the success of the ablation procedure Relationship between the location of LA low voltage areas and the success of the ablation procedure

CONTACTS AND LOCATIONS:
Overall Officials: Augustin Bortone, MD, Study Director — Elsan
Locations (13):
- France (13):
  - Infirmerie Protestante, Caluire-et-Cuire
  - CH Libourne, Libourne
  - CHU Lille, Lille
  - Hopital ST Phillbert, Lomme
  - CMC Ambroise Paré Hartmann, Neuilly-sur-Seine
  - Hôpital Privé Les Franciscaines, Nîmes
  - Hôpital Européen Georges Pompidou Service de cardiologie - Unité rythmologie, Paris
  - Clinique St Pierre Cardiologie, Perpignan
  - CHU Rennes, Rennes
  - CCN, Saint-Denis
  - Clinique Rhéna, Strasbourg
  - Clinique Pasteur Service de cardiologie/rythmologie, Toulouse
  - Chu Nancy, Vandœuvre-lès-Nancy

REFERENCES:
- [Background] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL. Corrigendum to: 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Oct 21;42(40):4194. doi: 10.1093/eurheartj/ehab648. No abstract available. PMID 34520521
- [Background] Verma A, Jiang CY, Betts TR, Chen J, Deisenhofer I, Mantovan R, Macle L, Morillo CA, Haverkamp W, Weerasooriya R, Albenque JP, Nardi S, Menardi E, Novak P, Sanders P; STAR AF II Investigators. Approaches to catheter ablation for persistent atrial fibrillation. N Engl J Med. 2015 May 7;372(19):1812-22. doi: 10.1056/NEJMoa1408288. PMID 25946280
- [Background] Sanders P, Hocini M, Jais P, Sacher F, Hsu LF, Takahashi Y, Rotter M, Rostock T, Nalliah CJ, Clementy J, Haissaguerre M. Complete isolation of the pulmonary veins and posterior left atrium in chronic atrial fibrillation. Long-term clinical outcome. Eur Heart J. 2007 Aug;28(15):1862-71. doi: 10.1093/eurheartj/ehl548. PMID 17341503
- [Background] Knecht S, Hocini M, Wright M, Lellouche N, O'Neill MD, Matsuo S, Nault I, Chauhan VS, Makati KJ, Bevilacqua M, Lim KT, Sacher F, Deplagne A, Derval N, Bordachar P, Jais P, Clementy J, Haissaguerre M. Left atrial linear lesions are required for successful treatment of persistent atrial fibrillation. Eur Heart J. 2008 Oct;29(19):2359-66. doi: 10.1093/eurheartj/ehn302. Epub 2008 Jul 8. PMID 18614522
- [Background] Valderrabano M, Peterson LE, Bunge R, Prystash M, Dave AS, Nagueh S, Kleiman NS. Vein of Marshall ethanol infusion for persistent atrial fibrillation: VENUS and MARS clinical trial design. Am Heart J. 2019 Sep;215:52-61. doi: 10.1016/j.ahj.2019.04.022. Epub 2019 May 11. PMID 31279972
- [Background] Kim DT, Lai AC, Hwang C, Fan LT, Karagueuzian HS, Chen PS, Fishbein MC. The ligament of Marshall: a structural analysis in human hearts with implications for atrial arrhythmias. J Am Coll Cardiol. 2000 Oct;36(4):1324-7. doi: 10.1016/s0735-1097(00)00819-6. PMID 11028490
- [Background] Valderrabano M, Chen HR, Sidhu J, Rao L, Ling Y, Khoury DS. Retrograde ethanol infusion in the vein of Marshall: regional left atrial ablation, vagal denervation and feasibility in humans. Circ Arrhythm Electrophysiol. 2009 Feb;2(1):50-6. doi: 10.1161/CIRCEP.108.818427. PMID 19756206
- [Background] Dave AS, Baez-Escudero JL, Sasaridis C, Hong TE, Rami T, Valderrabano M. Role of the vein of Marshall in atrial fibrillation recurrences after catheter ablation: therapeutic effect of ethanol infusion. J Cardiovasc Electrophysiol. 2012 Jun;23(6):583-91. doi: 10.1111/j.1540-8167.2011.02268.x. Epub 2012 Mar 19. PMID 22429895
- [Result] Pambrun T, Denis A, Duchateau J, Sacher F, Hocini M, Jais P, Haissaguerre M, Derval N. MARSHALL bundles elimination, Pulmonary veins isolation and Lines completion for ANatomical ablation of persistent atrial fibrillation: MARSHALL-PLAN case series. J Cardiovasc Electrophysiol. 2019 Jan;30(1):7-15. doi: 10.1111/jce.13797. Epub 2018 Dec 21. PMID 30461121
- [Result] Rivard L, Hocini M, Rostock T, Cauchemez B, Forclaz A, Jadidi AS, Linton N, Nault I, Miyazaki S, Liu X, Xhaet O, Shah A, Sacher F, Derval N, Jais P, Khairy P, Macle L, Nattel S, Willems S, Haissaguerre M. Improved outcome following restoration of sinus rhythm prior to catheter ablation of persistent atrial fibrillation: a comparative multicenter study. Heart Rhythm. 2012 Jul;9(7):1025-30. doi: 10.1016/j.hrthm.2012.02.016. Epub 2012 Feb 15. PMID 22342863
- [Result] Boveda S, Metzner A, Nguyen DQ, Chun KRJ, Goehl K, Noelker G, Deharo JC, Andrikopoulos G, Dahme T, Lellouche N, Defaye P. Single-Procedure Outcomes and Quality-of-Life Improvement 12 Months Post-Cryoballoon Ablation in Persistent Atrial Fibrillation: Results From the Multicenter CRYO4PERSISTENT AF Trial. JACC Clin Electrophysiol. 2018 Nov;4(11):1440-1447. doi: 10.1016/j.jacep.2018.07.007. Epub 2018 Aug 25. PMID 30466850
- [Result] Su WW, Reddy VY, Bhasin K, Champagne J, Sangrigoli RM, Braegelmann KM, Kueffer FJ, Novak P, Gupta SK, Yamane T, Calkins H; STOP Persistent AF Investigators. Cryoballoon ablation of pulmonary veins for persistent atrial fibrillation: Results from the multicenter STOP Persistent AF trial. Heart Rhythm. 2020 Nov;17(11):1841-1847. doi: 10.1016/j.hrthm.2020.06.020. Epub 2020 Jun 24. PMID 32590151
- [Result] Derval N, Duchateau J, Denis A, Ramirez FD, Mahida S, Andre C, Krisai P, Nakatani Y, Kitamura T, Takigawa M, Chauvel R, Tixier R, Pillois X, Sacher F, Hocini M, Haissaguerre M, Jais P, Pambrun T. Marshall bundle elimination, Pulmonary vein isolation, and Line completion for ANatomical ablation of persistent atrial fibrillation (Marshall-PLAN): Prospective, single-center study. Heart Rhythm. 2021 Apr;18(4):529-537. doi: 10.1016/j.hrthm.2020.12.023. Epub 2020 Dec 29. PMID 33383226
- [Derived] Bortone AA, Marijon E, Limite LR, Lagrange P, Brigadeau F, Martins R, Durand C, Albenque JP; PACIFIC study group. Pulmonary vein isolation alone or in combination with substrate modulation after electrical cardioversion failure in patients with persistent atrial fibrillation: The PACIFIC trial: Study design. J Cardiovasc Electrophysiol. 2023 Feb;34(2):270-278. doi: 10.1111/jce.15761. Epub 2022 Dec 7. PMID 36434797